CLINICAL TRIAL: NCT01319136
Title: Novel Infusion Method for Describing CSF Dynamics
Brief Title: Improved Analysis Methods for Infusion Tests
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Kennet Andersson, MSc, Umeå University
Other Study IDs: Dnr 08-130M
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2009-03

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: new infusion test method; reference method; cerebrospinal fluid dynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: Patients with Idiopathic Normal Pressure Hydrocephalus are improved with shunt surgery. To increase the accuracy of the diagnosis, supplementary tests that characterize the cerebrospinal fluid (CSF) dynamics are used. The infusion test is one of these, used for shunt surgery selection and postoperative evaluation of shunt function. Forty-eight patients that had a preoperative investigation because of communicating hydrocephalus at the university hospitals in Umeå and Uppsala, Sweden, participated in the study. The purpose of this study was to evaluate a new method, with a new infusion protocol and new analysis methods, and compare it to the current method.

ELIGIBILITY:
Inclusion Criteria:

* preoperative investigation because of communicating hydrocephalus
* ventriculomegaly (Evans ratio > 0.3)
* no obstruction to CSF flow at visual inspection

Exclusion Criteria:

* postoperative infusion test investigations
* patients that were unable to understand instructions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that had a preoperative investigation because of communicating hydrocephalus. MRI revealed ventriculomegaly (Evans ratio > 0.3), no obstruction to CSF flow at visual inspection. Most, but not all, fulfilled the criteria of "probable" or "possible" INPH.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Malm, PhD, MD, Study Director — Department of Clinical Neuroscience
Locations (2):
- Sweden (2):
  - Uppsala University Hospital, Uppsala, Uppland
  - Umeå University Hospital, Umeå, Västerbotten County